CLINICAL TRIAL: NCT00877474
Title: Phase I, Multicenter, Open-label, Dose-escalating, Clinical and Pharmacokinetic Study of PM01183 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-001-08
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: ADVANCED SOLID TUMORS
Keywords: PM01183; Solid tumors; PharmaMar USA
MeSH Terms: interventions — PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): PM01183 administered i.v. over one hour, on Day 1, every three weeks, at a starting dose of 20 µg/m2.
  Interventions: Drug: PM01183

INTERVENTIONS:
Drug: PM01183 — Vials containing 0.2 mg of PM01183 as powder for concentrate for solution for infusion

SUMMARY:
This is a phase I, multicenter, open-label, dose escalating clinical and pharmacokinetic study of PM01183 for patients with advanced solid tumors

DETAILED DESCRIPTION:
This is a phase I, multicenter, open-label, dose escalating clinical and pharmacokinetic study of PM01183 for patients with advanced solid tumors to identify the dose limiting toxicities (DLTs), determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 administered every three weeks intravenously (i.v.) over one hour to patients with advanced solid tumors and to preliminarily determine the pharmacokinetics of PM01183, to evaluate the antitumor activity of PM01183 and the safety and tolerability of PM01183. Besides this study will evaluate the pharmacogenomics in tumor samples and peripheral white blood cells (PWBCs) of patients exposed to PM01183 at the RD in order to assess potential markers of response and/or resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the patient obtained before any study-specific procedure.
2. Patients with histologically/cytologically confirmed diagnosis of advanced solid tumors refractory to standard therapy or for whom no standard therapy exist (excluding primary central nervous system tumors).
3. Age ≥ 18 years.
4. Patients with measurable or non-measurable disease according to RECIST.
5. Patients entered at the expansion cohort of the RD must have:

   * Measurable disease according to RECIST and/or, evaluable disease by serum markers in the case of prostate and ovarian cancer [according to the Prostate-Specific Antigen Working Group Recommendations (PSAWGR) and the Gynecologic Cancer Intergroup (GCIG) specific criteria, respectively].
   * Confirmed progressive disease after last therapy, before study initiation.
   * Available tumor samples (if pharmacogenomic study consented).
6. Recovery from any drug-related adverse event derived from any previous treatment, excluding alopecia and grade ≤ 1 asymptomatic peripheral neuropathy according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.3.0.
7. Laboratory values within seven days prior to first infusion:

   * Platelet count ≥ 100 x109/l, hemoglobin > 9 g/dl (patients can be transfused as clinically indicated prior to study entry) and absolute neutrophils count (ANC) ≥ 1.5 x109/l.
   * Alkaline phosphatase ≤ 2.5 x the upper limit of normality (ULN)
   * Aspartate aminotransferase (AST) ≤ 2.5 x ULN.
   * Alanine aminotransferase (ALT) ≤ 2.5 x ULN.
   * Total bilirubin ≤ ULN. f) Calculated creatinine clearance: ≥ 40 ml/min (calculated using the Cockcroft and Gault formula).
   * Albumin ≥ 2.5 g/dl.
   * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
8. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both men and women must agree to use a medically acceptable method of contraception throughout the treatment period and for 6 months after discontinuation of treatment. Acceptable methods of contraception include: intrauterine conceptive device (IUD), oral contraceptives, subdermal implant and double barrier (condom with a contraceptive sponge or contraceptive suppository).

Exclusion Criteria:

1. Pregnant or lactating women.
2. Less than three weeks from radiation therapy (six weeks in case of extensive prior radiotherapy) or last dose of hormonal therapy, biological therapy or chemotherapy (six weeks in case of nitrosoureas, mitomycin C, trastuzumab, bicalutamide or high-dose chemotherapy).
3. Evidence of progressive Central Nervous System (CNS) metastases or any symptomatic brain or leptomeningeal metastases.
4. Patients for whom non-standard surgery approach may result in tumor free survival or significant palliation.
5. Other relevant diseases or adverse clinical conditions:

   * Increased cardiac risk: symptomatic and/or medication requiring congestive heart failure or clinically relevant valvular heart disease or unstable angor pectoris or myocardial infarction within 12 months before inclusion in the study, or ≥ grade 1 arrhythmia or any grade requiring treatment, or uncontrolled arterial hypertension (≥ 160/100 mmHg) despite optimal medical therapy.
   * History of significant neurological or psychiatric disorders.
   * Active infection.
   * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
   * Immunocompromised patients, including those known to be infected by human immunodeficiency virus (HIV).
   * Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
6. Limitation of the patient's ability to comply with the treatment or to follow-up at a participating protocol. Patients registered on this trial must be treated and followed at a participating center.
7. Prior treatment with any investigational product in the period ≥ 5 half-lives of the investigational compound prior to the first infusion.
8. Known hypersensitivity to any of the components of the drug product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To identify the dose limiting toxicities (DLTs), determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 administered every three weeks intravenously (i.v.) over one hour to patients with advanced solid tumors. | Along the study

SECONDARY OUTCOMES:
To preliminarily determine: pharmacokinetics, antitumor activity and safety of PM01183 and to determine pharmacogenomics in tumor samples and peripheral white blood cells (PWBCs) at the RD | Along the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ratain, MD, Principal Investigator — Cancer Research Center. University of Chicago Hospitals.; Josep Tabernero, MD, Principal Investigator — Vall d'Hebron University Hospital. Barcelona (Spain)
Locations (2):
- Cancer Research Center. University of Chicago Hospitals., Chicago, Illinois, United States
- Vall d'Hebron University Hospital., Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Fernandez-Teruel C, Lubomirov R, Fudio S. Population Pharmacokinetic-Pharmacodynamic Modeling and Covariate Analyses of Neutropenia and Thrombocytopenia in Patients With Solid Tumors Treated With Lurbinectedin. J Clin Pharmacol. 2021 Sep;61(9):1206-1219. doi: 10.1002/jcph.1886. Epub 2021 Jun 9. PMID 33914350
- [Derived] Elez ME, Tabernero J, Geary D, Macarulla T, Kang SP, Kahatt C, Pita AS, Teruel CF, Siguero M, Cullell-Young M, Szyldergemajn S, Ratain MJ. First-in-human phase I study of Lurbinectedin (PM01183) in patients with advanced solid tumors. Clin Cancer Res. 2014 Apr 15;20(8):2205-14. doi: 10.1158/1078-0432.CCR-13-1880. Epub 2014 Feb 21. PMID 24563480